CLINICAL TRIAL: NCT00174252
Title: Evolution of IGF-1 in Children Born Small for Gestational Age and With Growth Retardation, Treated by Genotonorm Especially Evolution After Dose Adaptation.
Brief Title: Study Aimed At Improving Height With Genotonorm In Children Born Little And/Or Light With Growth Retardation At The Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6281234
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Results first posted 2010-06-04 (Estimated); Last update posted 2010-06-15 (Estimated); Status verified 2009-06

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genotonorm (Somatropin) (Experimental)
  Interventions: Drug: Genotonorm (Somatropin)

INTERVENTIONS:
Drug: Genotonorm (Somatropin) — 0.40 mg/kg/week dived in 7 daily subcutaneous injections during 2 years

SUMMARY:
To estimate the percentage of children with serum IGF-1 > 2 standard deviation (compared to a child of the same gender and age and without growth hormone (GH) deficiency) 9 months and 12 months after initiation of GH treatment.

ELIGIBILITY:
Inclusion Criteria:

* Chronological age between 4 and 9 years for a boy and 4 and 7 years for a girl.
* Measured Height < -2.5 Standard Deviation

Exclusion Criteria:

* Pubertal signs ie: testis volume > or = 4 ml in boys and breast stage > or = B2 (Tanner)
* Serious chronic disease (diabetes, renal insufficiency, heart failure, hepatic insufficiency, neoplasia)

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2005-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- France (19):
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Besançon
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Bron
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Dunkirk
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Limoges
  - Pfizer Investigational Site, Lorient
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Rennes
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Tarbes
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Tours
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6281234&StudyName=Study%20Aimed%20At%20Improving%20Height%20With%20Genotonorm%20In%20Children%20Born%20Little%20And/Or%20Light%20With%20Growth%20Retardation%20At%20The%20Age

RESULTS

PARTICIPANT FLOW:
Groups:
- Genotonorm: Initiated at a dose of 0.40 milligrams (mg)/kilograms (kg) of Genotonorm divided in 7 daily subcutaneous injections and titrated as needed.
Period: Overall Study
Arm/Group | Genotonorm
Started | 57
Completed | 55
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Genotonorm
Number analyzed (Participants) | 57
Age, Customized [Number; unit: participants]
  <4 years | 1
  Between 4 and 8 years | 49
  Between 8 and 12 years | 7
  >=12 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 23

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Change in Height From Baseline
Description: The standing height measurements were performed at the same time of the day by using a wallmounted device (e.g. Harpenden Stadiometer) at each study visit. The pre-specified clinical outcomes were analyzed at 12 and 24 months.
Time Frame: Baseline, 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children with evaluable height data at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Genotonorm
Number analyzed (Participants) | 55
centimeters (cm)
  12 Months | 9.0 (1.3)
  24 Months | 16.4 (2.2)

2. Primary Outcome: Percentage of Children With Insulin Growth Factor-1 (IGF-1) > 2 Standard Deviation (SD) at 9 and 12 Months
Description: Percentage of children with serum IGF-1 > 2 SD (compared to a child of the same gender and age and without growth hormone (GH) deficiency) 9 months and 12 months after initiation of GH treatment. 9 months and 12 months are combined.
Time Frame: 9 and 12 months
Population: The safety analysis set (SAS) was defined as all patients who received at least one dose of GH treatment. Number of Participants Analyzed = Number of children treated.
Measure: Number; unit: percentage of participants
Arm/Group | Genotonorm
Number analyzed (Participants) | 57
percentage of participants
  No | 86.0
  Yes | 14.0
Statistical Analysis 1: Comparison: Genotonorm; Applies to "no"; Test type: Superiority or Other; Percentage = 86.0, 95% CI 2-sided [74.2 to 93.7] — 95% CI was estimated using the F-distribution
Statistical Analysis 2: Comparison: Genotonorm; Applies to "yes"; Test type: Superiority or Other; Percentage = 14.0, 95% CI [6.3 to 25.8] — 95% confidence interval (CI) was estimated using the F-distribution

3. Secondary Outcome: Change in Height SD Chronological Age (CA) From Baseline at 12 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months
Description: The height in SD was calculated using Sempe reference means and standard deviations for height. Change in height SD was calculated as height in SD at "12 months" minus height in SD at "Baseline".
Time Frame: Baseline, 12 months
Population: The full analysis set (FAS) included all patients who received at least one dose of assigned treatment and had at least one subsequent rating of IGF-1. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable height SD CA data at 12 months.
Measure: Mean (Standard Deviation); unit: SD for CA
Arm/Group | Genotonorm
Number analyzed (Participants) | 46
SD for CA | 0.81 (0.26)

4. Secondary Outcome: Change in Height SD CA From Baseline at 24 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months
Description: The height in SD was calculated using Sempe reference means and SDs for height. Change in height SD was calculated as height in SD at "24 months" minus height in SD at "Baseline".
Time Frame: Baseline, 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable height SD CA data at 24 months.
Measure: Mean (Standard Deviation); unit: SD for CA
Arm/Group | Genotonorm
Number analyzed (Participants) | 47
SD for CA | 1.24 (0.48)

5. Secondary Outcome: Change in Height SD CA From Baseline at 12 and 24 Months in Children With IGF-1 > 2 SD at 9 and 12 Months
Description: The height in SD was calculated using Sempe reference means and SDs for height. Change in height SD was calculated as height in SD at "12 or 24 months" minus height in SD at "Baseline".
Time Frame: Baseline, 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 > 2 SD at 9 and 12 months with evaluable Height SD CA data at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: SD for BA
Arm/Group | Genotonorm
Number analyzed (Participants) | 8
SD for BA
  12 Months | 1.13 (0.35)
  24 Months | 1.53 (0.20)

6. Secondary Outcome: Change in Height SD Bone Age (BA) From Baseline at 12 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months
Description: The height in SD was calculated using Sempe reference means and SDs for height. Change in height SD was calculated as height in SD at "12 months" minus height in SD at "Baseline".
Time Frame: Baseline, 12 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable height SD BA data at 12 months.
Measure: Mean (Standard Deviation); unit: SD for BA
Arm/Group | Genotonorm
Number analyzed (Participants) | 33
SD for BA | 0.44 (1.34)

7. Secondary Outcome: Change in Height SD BA From Baseline at 24 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months
Description: as for outcome 4
Time Frame: Baseline, 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable height SD BA data at 24 months.
Measure: Mean (Standard Deviation); unit: Height in SD
Arm/Group | Genotonorm
Number analyzed (Participants) | 31
Height in SD | 0.12 (1.86)

8. Secondary Outcome: Change in Height SD BA From Baseline at 12 and 24 Months in Children With IGF-1 > 2 SD at 9 and 12 Months
Description: as for outcome 5
Time Frame: Baseline, 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 > 2 SD at 9 or 12 months with evaluable height SD BA data at 12 and 12 months.
Measure: Mean (Standard Deviation); unit: SD for BA
Arm/Group | Genotonorm
Number analyzed (Participants) | 7
SD for BA
  12 Months | 0.64 (1.19)
  24 Months | 0.64 (1.30)

9. Other Pre Specified Outcome: Growth Rate at 12 and 24 Months
Description: Growth Rate was calculated at 12 months as:
  (Height at 12 months minus Height at Day 0) divided by {(Date of 12 months minus Date of Day 0) divided by 365.25}
  Growth Rate was calculated at 24 months as:
  (Height at 24 months minus Height at 12 months) divided by {(Date of 24 months minus Date of 12 months) divided by 365.25}
Time Frame: 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children treated. n = Number of children with evaluable growth rate data at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Genotonorm
Number analyzed (Participants) | 57
cm/year
  12 Months | 9.06 (1.40)
  24 Months (n=55) | 7.23 (1.38)

10. Secondary Outcome: Summary of Growth Rate SD (CA) at 12 and 24 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months
Description: Growth rate SD CA at 12 months was calculated as:(Growth rate at 12 months minus reference mean for CA at 12 months) divided by reference SD for CA at 12 months
  Growth rate SD CA at 24 months was calculated as:(Growth rate at 24 months minus reference mean for CA at 24 months) divided by reference SD for CA at 24 months
Time Frame: 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable growth rate SD CA data at 12 months. n = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable growth rate SD CA data at 24 months.
Measure: Mean (Standard Deviation); unit: SD for CA
Arm/Group | Genotonorm
Number analyzed (Participants) | 49
SD for CA
  12 Months | 3.77 (1.68)
  24 Months (n=47) | 1.74 (1.51)

11. Secondary Outcome: Summary of Growth Rate SD (CA) at 12 and 24 Months in Children With IGF-1 > 2 SD at 9 and 12 Months
Description: Growth rate SD CA at 12 months was calculated as: (Growth rate at 12 months minus reference mean for CA at 12 months) divided by reference SD for CA at 12 months
  Growth rate SD CA at 24 months was calculated as: (Growth rate at 24 months minus reference mean for CA at 24 months) divided by reference SD for CA at 24 months
Time Frame: 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 > 2 SD at 9 and 12 months with evaluable growth rate SD CA data at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: SD for CA
Arm/Group | Genotonorm
Number analyzed (Participants) | 8
SD for CA
  12 Months | 5.24 (1.64)
  24 Months | 2.15 (2.21)

12. Secondary Outcome: Summary of Growth Rate SD (BA) at 12 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months
Description: Growth rate SD BA at 12 months was calculated as: (Growth rate at 12 months minus reference mean for BA at 12 months) divided by reference SD for BA at 12 months
Time Frame: Baseline, 12 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable growth rate SD BA data at 12 months.
Measure: Mean (Standard Deviation); unit: SD for CA
Arm/Group | Genotonorm
Number analyzed (Participants) | 33
SD for CA | 2.38 (1.88)

13. Secondary Outcome: Summary of Growth Rate SD (BA) at 24 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months
Description: Growth rate SD BA at 24 months was calculated as: (Growth rate at 24 months minus reference mean for BA at 24 months) divided by reference SD for BA at 24 months
Time Frame: Baseline, 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable growth rate SD BA data at 24 months.
Measure: Mean (Standard Deviation); unit: SD for BA
Arm/Group | Genotonorm
Number analyzed (Participants) | 39
SD for BA | 1.26 (1.62)

14. Secondary Outcome: Summary of Growth Rate SD (BA) at 12 and 24 Months in Children With IGF-1 > 2 SD at 9 and 12 Months
Description: Growth rate SD BA at 12 months was calculated as: (Growth rate at 12 months minus reference mean for BA at 12 months) divided by reference SD for CA at 12 months
  Growth rate SD BA at 24 months was calculated as: (Growth rate at 24 months minus reference mean for BA at 24 months) divided by reference SD for CA at 24 months
Time Frame: 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 > 2 SD at 9 and 12 months with evaluable growth rate SD BA data at 12 months. n = Number of children with IGF-1 > 2 SD at 9 and 12 months with evaluable growth rate SD BA data at 24 months.
Measure: Mean (Standard Deviation); unit: SD for BA
Arm/Group | Genotonorm
Number analyzed (Participants) | 7
SD for BA
  12 Months | 4.02 (2.37)
  24 Months (n=6) | 1.71 (2.26)

15. Other Pre Specified Outcome: Summary of Body Mass Index (BMI) at 12 and 24 Months
Description: BMI was calculated at 12 months and 24 months as: (Weight at 12 or 24 months divided by Height at 12 or 24 months) squared
Time Frame: 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children treated. n = Number of children with evaluable BMI data at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: kg/meters squared (m2)
Arm/Group | Genotonorm
Number analyzed (Participants) | 57
kg/meters squared (m2)
  12 Months (n=54) | 14.7 (1.5)
  24 Months (n=55) | 14.9 (1.4)

16. Secondary Outcome: Analysis of Covariance (ANCOVA) for Height SD CA at 12 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months and IGF-1 > 2 SD at 9 and 12 Months
Description: Change in Height SD (CA) was calculated as:
  Height SD (CA) at 12 months minus Height SD (CA) at Baseline
Time Frame: Baseline, 12 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months or with IGF-1 > 2 SD at 9 and 12 months and with evaluable height SD CA data at 12 months.
Measure: Mean (Standard Error); unit: SD for CA
Arm/Group | Genotonorm (IGF-1 < = 2 SD at 9 or 12 Months) | Genotonorm (IGF-1 > 2 SD at 9 and 12 Months)
Number analyzed (Participants) | 46 | 8
SD for CA | -1.94 (0.04) | -1.59 (0.10)
Statistical Analysis 1: Comparison: Genotonorm (IGF-1 < = 2 SD at 9 or 12 Months) vs Genotonorm (IGF-1 > 2 SD at 9 and 12 Months); Test type: Superiority or Other; p = 0.002, ANCOVA; Adjusted for height SD at baseline; Mean Difference (Net) = -0.35

17. Secondary Outcome: ANCOVA for Height SD CA at 24 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months and IGF-1 > 2 SD at 9 and 12 Months
Description: Height SD (CA) at 24 months.
Time Frame: Baseline, 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months or with IGF-1 > 2 SD at 9 and 12 months and with evaluable height SD CA data at 24 months.
Measure: Mean (Standard Error); unit: SD for CA
Arm/Group | Genotonorm (IGF-1 < = 2 SD at 9 or 12 Months) | Genotonorm (IGF-1 > 2 SD at 9 and 12 Months)
Number analyzed (Participants) | 44 | 8
SD for CA | -1.53 (0.06) | -1.18 (0.14)
Statistical Analysis 1: Comparison: Genotonorm (IGF-1 < = 2 SD at 9 or 12 Months) vs Genotonorm (IGF-1 > 2 SD at 9 and 12 Months); Test type: Superiority or Other; p = 0.023, ANCOVA — Bilateral test multiple comparison threshold for statistical significance = 0.05; Adjusted for height SD at baseline; Mean Difference (Net) = -0.35

18. Secondary Outcome: ANCOVA for Height SD BA at 12 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months and IGF-1 > 2 SD at 9 and 12 Months
Description: Change in Height SD (BA) was calculated as:
  Height SD (BA) at 12 months minus Height SD (BA) at Baseline
Time Frame: Baseline, 12 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months or with IGF-1 > 2 SD at 9 and 12 months and with evaluable height SD BA data at 12 months.
Measure: Mean (Standard Error); unit: SD for BA
Arm/Group | Genotonorm (IGF-1 < = 2 SD at 9 or 12 Months) | Genotonorm (IGF-1 > 2 SD at 9 and 12 Months)
Number analyzed (Participants) | 33 | 7
SD for BA | 0.56 (0.22) | 0.76 (0.48)
Statistical Analysis 1: Comparison: Genotonorm (IGF-1 < = 2 SD at 9 or 12 Months) vs Genotonorm (IGF-1 > 2 SD at 9 and 12 Months); Test type: Superiority or Other; p = 0.708, ANCOVA; Adjusted for height SD at baseline; Mean Difference (Final Values) = -0.20

19. Secondary Outcome: ANCOVA for Height SD BA at 24 Months in Children With IGF-1 <= 2 SD at 9 or 12 Months and IGF-1 > 2 SD at 9 and 12 Months
Description: Height SD (BA) at 24 months
Time Frame: Baseline, 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months or with IGF-1 > 2 SD at 9 and 12 months and with evaluable height SD BA data at 24 months.
Measure: Mean (Standard Error); unit: SD for BA
Arm/Group | Genotonorm (IGF-1 < = 2 SD at 9 or 12 Months) | Genotonorm (IGF-1 > 2 SD at 9 and 12 Months)
Number analyzed (Participants) | 31 | 7
SD for BA | 0.05 (0.25) | 0.64 (0.53)
Statistical Analysis 1: Comparison: Genotonorm (IGF-1 < = 2 SD at 9 or 12 Months) vs Genotonorm (IGF-1 > 2 SD at 9 and 12 Months); Test type: Superiority or Other; p = 0.325, ANCOVA; Adjusted for height SD at baseline; Mean Difference (Net) = -0.59

20. Other Pre Specified Outcome: Change in BA From Baseline at 12 and 24 Months
Description: Change in BA was calculated as: (12 or 24 months minus Screening)
Time Frame: Baseline, 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children treated. n = Number of children with evaluable BA data at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: year
Arm/Group | Genotonorm
Number analyzed (Participants) | 57
year
  12 Months (n=33) | 1.2 (0.9)
  24 Months (n=31) | 2.5 (1.1)

21. Other Pre Specified Outcome: BA/CA at 12 and 24 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months
Description: The BA/CA ratio was calculated at Screening, 12 and 24 months. The CA was the age on the date that the corresponding BA X-ray was performed.
Time Frame: 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable BA/CA data at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Genotonorm
Number analyzed (Participants) | 43
ratio
  12 Months | 0.74 (0.17)
  24 Months | 0.82 (0.16)

22. Other Pre Specified Outcome: BA/CA at 12 and 24 Months in Children With IGF-1 > 2 SD at 9 and 12 Months
Description: as for outcome 21
Time Frame: 12 and 24 months
Population: FAS. Number of Participants Analyzed = Number of children with IGF-1 > 2 SD at 9 and 12 months with evaluable BA/CA data at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Genotonorm
Number analyzed (Participants) | 7
ratio
  12 Months | 0.80 (0.21)
  24 Months | 0.83 (0.09)

23. Secondary Outcome: Summary of IGF-1 SD at 6, 9, 12, 15, 18, 21, and 24 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months
Description: IGF-1 SD was calculated at each study time point using gender specific IGF-1 reference mean and SD for the CA of the child on the date of the corresponding IGF-1 blood sample: IGF-1 SD = (IGF-1 minus reference mean) divided by reference SD
Time Frame: 6, 9, 12, 15, 18, 21, and 24 months
Population: SAS. Number of Participants Analyzed = Number of children treated. n = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable IGF-1 SD data at 6, 9, 12, 15, 18, 21, and 24 months.
Measure: Mean (Standard Deviation); unit: SD
Arm/Group | Genotonorm
Number analyzed (Participants) | 57
SD
  6 Months (n=49) | 0.65 (1.11)
  9 Months (n=46) | 0.93 (1.26)
  12 Months (n=44) | 1.04 (0.96)
  15 Months (n=40) | 0.88 (1.28)
  18 Months (n=43) | 0.88 (1.17)
  21 Months (n=41) | 0.82 (0.93)
  24 Months (n=45) | 0.85 (1.17)

24. Secondary Outcome: Summary of IGF-1 SD at 6, 9, 12, 15, 18, 21, and 24 Months in Children With IGF-1 > 2 SD at 9 and 12 Months
Description: IGF-1 SD was calculated at each study time point using these gender specific IGF-1 reference means and SDs for the CA of the child on the date of the corresponding IGF-1 blood sample: IGF-1 SD = (IGF-1 - reference mean) / reference SD
Time Frame: 6, 9, 12, 15, 18, 21, and 24 months
Population: SAS. Number of Participants Analyzed = Number of children treated. n = Number of children with IGF-1 > 2 SD at 9 and 12 months with evaluable IGF-1 SD data at 6, 9, 12, 15, 18, 21, and 24 months.
Measure: Mean (Standard Deviation); unit: SD
Arm/Group | Genotonorm
Number analyzed (Participants) | 57
SD
  6 Months (n=7) | 2.32 (0.68)
  9 Months (n=6) | 2.35 (0.19)
  12 Months (n=8) | 2.50 (0.27)
  15 Months (n=7) | 1.40 (1.08)
  18 Months (n=7) | 2.12 (1.18)
  21 Months (n=7) | 1.82 (1.09)
  24 Months (n=8) | 1.81 (1.03)

25. Secondary Outcome: IGF-1/Insulin-Like Growth Factor Binding Protein 3 (IGFBP-3) Ratio at 12 and 24 Months in Children With IGF-1 < = 2 SD at 9 or 12 Months
Time Frame: 12 and 24 months
Population: SAS. Number of Participants Analyzed = Number of children treated. n = Number of children with IGF-1 < = 2 SD at 9 or 12 months with evaluable IGF-1/IGFBP-3 data at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Genotonorm
Number analyzed (Participants) | 57
ratio
  12 Months (n=44) | 0.17 (0.06)
  24 Months (n=45) | 0.19 (0.07)

26. Secondary Outcome: IGF-1/IGFBP-3 Ratio at 12 and 24 Months in Children With IGF-1 > 2 SD at 9 and 12 Months
Time Frame: 12 and 24 months
Population: SAS. Number of Participants Analyzed = Number of children with IGF-1 > 2 SD at 9 and 12 months with evaluable IGF-1/IGFBP-3 data at 12 and 24 months.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Genotonorm
Number analyzed (Participants) | 8
ratio
  12 Months | 0.23 (0.03)
  24 Months | 0.21 (0.06)

ADVERSE EVENTS:
Arm/Group | Genotonorm
Serious Adverse Events (participants affected / at risk) | 6/57
Other Adverse Events (participants affected / at risk) | 30/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotonorm (N=57)
Amniotic band syndrome (Congenital, familial and genetic disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Pneumonia (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Genotonorm (N=57)
Microcytosis (Blood and lymphatic system disorders) | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Conjunctivitis (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Eyelid oedema (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
House dust allergy (Immune system disorders) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 5
Ear infection (Infections and infestations) | 3
Furuncle (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Influenza (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Lyme disease (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 4
Skin infection (Infections and infestations) | 1
Tinea infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 1
Varicella (Infections and infestations) | 6
Viral infection (Infections and infestations) | 1
Vulvitis (Infections and infestations) | 1
Insulin-like growth factor increased (Investigations) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 5
Sleep disorder (Psychiatric disorders) | 1
Sleep terror (Psychiatric disorders) | 1
Enuresis (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Adenotonsillectomy (Surgical and medical procedures) | 1
Tonsillectomy (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.